CLINICAL TRIAL: NCT03552679
Title: A Prospective, Multicenter, Observational, Investigator Initiated Study, Aiming at Serial Multiparametric Evaluation of Right Ventricular Function to Predict Optimal Management Strategies, of Right Heart Failure After LVAD Implantation
Brief Title: Serial Multiparametric Evaluation of Right Ventricular Function After Left Ventricular Assist Device Implantation
Acronym: EuroEchoVAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: The European Association for Cardio-Thoracic Surgery (Unknown)
Responsible Party: Principal Investigator, I. Osama SOLIMAN, Assistant Professor of Cardiology, Erasmus Medical Center
Other Study IDs: WT/aj/MEC-2018-1162
Record Dates: First submitted 2018-05-27; First posted 2018-06-12 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Right Heart Failure
Keywords: Right Heart Failure; Ventricular Assist Device; Mortality; ICU Stay; Acute Kidney Injury
MeSH Terms: conditions — Heart Failure; Acute Kidney Injury | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LVAD recipients: Consecutive patients accepted for elective LVAD implantation in the context of routine care, will undergo routinely scheduled echocardiography before, within 1 week, 1 month, 3 months and 1 year after LVAD implantation. Echocardiography will be performed using ultrasound machines that are capable of acquisition of two-, three-dimensional and Multiplane Echocardiography of the right ventricle. Invasive hemodynamic data will be collected in the perioperative period.
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography

SUMMARY:
The primary purpose of this study is to investigate the evolution of Right Ventricular (RV) function before and after left ventricular assist device (LVAD) implantation, using novel echocardiographic quantification of RV size and function in combination with comprehensive hemodynamic, laboratory and clinical parameters. The findings of the study will enhance prediction of early and late development of postoperative right-sided heart failure (RHF) and subsequent mortality and morbidity.

The secondary purpose of the study is to combine echocardiographic, hemodynamic, laboratory, and clinical data to define optimal management strategies of RHF after LVAD implantation.

DETAILED DESCRIPTION:
The study consists of 2 parts: a Pilot study and a Main Study as detailed below.

The purpose of the Pilot study is to evaluate the feasibility of RV quantification using two-, three-dimensional and Multiplane echocardiography.

About 100 subjects undergoing LVAD implantation in the European Registry for Patients with Mechanical Circulatory Support (EUROMACS) Registry are included in the Pilot study. These 100 patients will undergo routinely scheduled echocardiography before, within 1 week, 3 months and 1 year after LVAD implantation. Echocardiography will be performed using ultrasound machines that are capable of acquisition of two-, three-dimensional and Multiplane Echocardiography of the right ventricle.

Echocardiographic analysis will include three-dimensional quantification of the RV size and function as well as RV strain analysis in the Multiplane format as described in the Appendix Echocardiography Procedure Manual.

The Echocardiographic analyses of the first 50 patients, included in selected sites, will be used to further specify the protocol for image acquisition and analysis to be used in the Main Study. Furthermore, all sites will first enter 2 patients in the Pilot Study before they can participate in the Main Study. The echocardiographic results of these 2 patients will be assessed by the core lab for quality.

The purpose of the Main Study is to assess the evolution of RV function before and after LVAD implantation utilizing the acquisition and analysis protocol developed in the Pilot Study.

500 patients will undergo routinely scheduled echocardiographic imaging before LVAD implantation, and at 1 week, 1 month, 3 months, 6 months and 1 year thereafter. Echocardiography will be performed using the detailed protocol developed in the Pilot Study. All Echocardiographic images will be submitted to an independent Core Laboratory for analysis.

The evolution of RV function will be documented with standardised two-, three-dimensional and Multiplane Echocardiography of the right ventricle. The echocardiographic parameters include: RV strain and strain rate, RV Fractional Area Change, RV longitudinal function, RV volumes, RV ejection fraction, tricuspid regurgitation severity, estimated pulmonary artery pressures, pulmonary artery resistance, pulmonary artery compliance, RV stroke work index, right atrial size, and RV - pulmonary coupling.

Invasive hemodynamic data will be collected in the perioperative period. These RV parameters will be linked to the occurrence of clinical signs, hemodynamic and laboratory evidence of RHF.

ELIGIBILITY:
Inclusion Criteria:

Subjects to be included in the study must meet the following inclusion criteria:

1. Consecutive patients accepted for elective LVAD implantation in the context of routine care
2. >17 years of age
3. Written informed consent (IC), either by the patient or by legal representatives
4. Treated with mainstream devices

Exclusion Criteria:

* None

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who underwent LVAD implantation using main stream devices
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-06-24 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Moderate or severe RHF | 12 months
  RHF is defined by a triad of:
  1. Clinical (right-sided congestion, with or without hypotension, or hypo-perfusion)
  2. Imaging evidence (RV dilatation, new > grade 2 tricuspid regurgitation) deterioration right ventricular function score assessed by the echocardiography core laboratory)
  3. Hemodynamic evidence (discordant elevated central venous pressure (CVP) or right atrial pressure (RAP) >16 mmHg, despite normal or steady pulmonary capillary wedge pressure (PCWP), or right atrial (RA) to PCWP ratio >0.54).

SECONDARY OUTCOMES:
Severe RHF composite | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of Severe RHF composite after LVAD implantation
All-cause death | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of all-cause death after LVAD implantation
Cardiovascular death | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of cardiovascular death after LVAD implantation
Death or urgent transplantation | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of death or urgent transplantation after LVAD implantation
Length of post-operative Intensive Care Unit (ICU) stay | 30 days, 90 days, 180 days, 12 months
  The length of post-operative ICU stay in days after LVAD implantation
Length of post-operative hospital stay | 30 days, 90 days, 180 days, 12 months
  The length of post-operative hospital stay in days after LVAD implantation
Readmissions for heart failure or RHF | 30 days, 90 days, 180 days, 12 months
  The occurrence of hospital readmissions for heart failure or RHF after LVAD implantation
Sepsis | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of sepsis after LVAD implantation
LVAD and driveline-related infection | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of LVAD and driveline-related infection after LVAD implantation
Early and late bleeding complications | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of LVAD and driveline-related infection after LVAD implantation
LVAD pump thrombosis | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of LVAD and driveline-related infection after LVAD implantation
Haemolysis | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of LVAD and driveline-related infection after LVAD implantation
Arterial thromboembolic events, including stroke | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of LVAD and driveline-related infection after LVAD implantation
Venous thromboembolic events, including deep venous thrombosis (DVT) and pulmonary embolism (PE) | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of LVAD and driveline-related infection after LVAD implantation
Ventricular arrhythmias, either sustained symptomatic or with appropriate Implantable Cardioverter Defibrillator (ICD) therapy | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of LVAD and driveline-related infection after LVAD implantation
Atrial arrhythmias - documented atrial flutter or fibrillation | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of LVAD and driveline-related infection after LVAD implantation
Acute Kidney Injury (AKI) according to Kidney Disease Outcomes Quality Initiative (KDIGO) and RIFFLE criteria | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of LVAD and driveline-related infection after LVAD implantation
Chronic kidney disease (CKD) according to KDOQI criteria | 1 week, 30 days, 90 days, 180 days, 12 months
  The occurrence of Chronic kidney disease (CKD) according to KDOQI criteria after LVAD implantation
Six Minute walk distance in meters | 90 days and 12 months
  Assessment of Six Minute walk distance in meters before and after LVAD implantation
Quality of life (QoL) scores | 90 days, 180 days and at 12 months
  QoL by multiple assessments before and at 90 days, 180 days and at 12 months after LVAD implantation at

CONTACTS AND LOCATIONS:
Overall Officials: Osama SOLIMAN, MD, PhD, Principal Investigator — Euro Heart Foundation; Kadir Caliskan, MD, PhD, Principal Investigator — Erasmus MC Rotterdam
Locations (9):
- Germany (2):
  - Herz- und Diabeteszentrum Nordrhein- Westfalen, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
- Heart Center of the Semmelweis University, Budapest, Hungary
- Italy (2):
  - S. Orsola Hospital, Bologna University, Bologna
  - Ospedale dei Colli, Naples
- National Research Cardiac Surgery Center, Astana, Kazakhstan
- Erasmus Medical Center, Rotterdam, Netherlands
- Ege University School of Medicine, Izmir, Turkey (Türkiye)
- Euromacs, Eacts, Windsor, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soliman OII, Akin S, Muslem R, Boersma E, Manintveld OC, Krabatsch T, Gummert JF, de By TMMH, Bogers AJJC, Zijlstra F, Mohacsi P, Caliskan K; EUROMACS Investigators. Derivation and Validation of a Novel Right-Sided Heart Failure Model After Implantation of Continuous Flow Left Ventricular Assist Devices: The EUROMACS (European Registry for Patients with Mechanical Circulatory Support) Right-Sided Heart Failure Risk Score. Circulation. 2018 Feb 27;137(9):891-906. doi: 10.1161/CIRCULATIONAHA.117.030543. Epub 2017 Aug 27. PMID 28847897